CLINICAL TRIAL: NCT04913740
Title: Nursing Study of Skin Lesions Related to Health Care Protection COVID-19 Epidemic
Brief Title: Nursing Study of Skin Lesions Related to Health Care Protection in Novel Nursing Study of Skin Lesions Related to Health Care Protection in Novel Coronavirus Epidemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2020-841
Record Dates: First submitted 2021-06-02; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Associated Skin Lesions
MeSH Terms: interventions — Ointments; Bandages

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): health care workers who did not use any preventive measures on the basis of tertiary protection
- Experimental group (Experimental): On the basis of three-level protection, skin correlation prevention is carried out:
  1. pay attention to the protection of exposed skin, so that it is local dry.
  2. Do a good job of facial moisturizing work before workuse moisturizing ointment, more durable and non-irritating cream or emulsion, such as vitamin E cream, petroleum jelly, to do a good job of moisturizing work.
  3. Use appropriate dressing to avoid direct contact between the mask and the skin, and select the appropriate type of protective device; Reduce friction by applying foam patches, hydrocolloidal dressings, and empleters to the hair area. However, it should be noted that it must be confirmed that airtightness is good and that the protective effect is still the primary purpose of the medical staff.
  4. After work, avoid using irritantsto clean the face, and massage local skin with skin moisturizer; (5) If severe skin damage occurs, treat it as prescribed by the doctor
  Interventions: Other: Ointment and dressing for external use

INTERVENTIONS:
Other: Ointment and dressing for external use — 1. pay attention to the protection of exposed skin, so that it is local dry.
  2. Do a good job of facial moisturizing work before work use moisturizing ointment, more durable and non-irritating cream or emulsion, such as vitamin E cream, petroleum jelly, to do a good job of moisturizing work.
  3. Use appropriate dressing to avoid direct contact between the mask and the skin, and select the appropriate type of protective device; Reduce friction by applying foam patches, hydrocolloidal dressings, and empleters to the hair area. However, it should be noted that it must be confirmed that airtightness is good and that the protective effect is still the primary purpose of the medical staff.
  4. After work, avoid using irritants to clean the face, and massage local skin with skin moisturizer; (5) If severe skin damage occurs, treat it as prescribed by the doctor
  Arms: Experimental group

SUMMARY:
In the fight against the epidemic, medical personnel need to wear protective equipment, such as N95 mask, face screen, goggles, latex gloves, waterproof isolation clothing, and have special requirements. Protection-related skin lesions after the use of protective equipment will affect the health and comfort of medical workers. In this study, a retrospective study was conducted on the front-line medical workers in the fight against COVID-19 using questionnaires, so as to understand the incidence, location and clinical manifestations of skin lesions caused by the use of protective equipment by medical workers. And analyze the causes of these skin damage, so as to develop the corresponding prevention and treatment countermeasures, select 170 cases that meet the research conditions, a randomized controlled experiment, divided into control group and experimental group: the control group is on the basis of three-level protection, did not use any preventive measures of health care workers. In the experimental group, skin related prevention was carried out on the basis of three-level protection. The specific interventions are as follows :(1) Focus on protecting exposed skin and making it locally dry. (2) Do a good job of facial moisturizing before work (at least 1 hour before wearing the mask), use moisturizing ointment, longer lasting and non-irritating cream or emulsion, such as vitamin E cream, Vaseline, avoid direct contact with the skin of the mask, choose the appropriate type of protective device; Reduce friction by sticking foam paste, hydrocolloid accessories, ampute and so on on good hair parts. However, it should be noted that it must be confirmed that the airtightness is good, and the primary purpose of the medical staff is to ensure the protective effect. (4) After work, avoid using irritant (such as hot water, exfoliating cream, etc.) to clean the face, and massage local skin with skin moisturizer; (5) In case of severe skin damage, treat as prescribed by the doctor; (6) After finishing the front-line work, "Questionnaire Star" was used to collect data, and all data were input into the statistical software for analysis to compare the index differences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Job post: fever clinic, COVID-19 throat swab sampling site, isolation ward
2. Health care workers who have worked for 30 days or more
3. The continuous working time of tertiary protection shall be more than or equal to 4 hours
4. Signed the informed consent and volunteered to participate in the study.

Exclusion Criteria:

1. Existing long-term skin damage
2. The skin damage related to protection is too heavy to be studied

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of skin damage caused by the use of protective equipment by health care workers | 1year

CONTACTS AND LOCATIONS:
Overall Officials: ZeXing Chen, Study Chair — supervision
Locations (1):
- Dressing, Hangzhou, Zhejiang, China